CLINICAL TRIAL: NCT02728479
Title: PTA Registry - an Observational Study of Percutaneous Transluminal Angioplasty
Brief Title: Percutaneous Transluminal Angioplasty Registry
Status: Recruiting | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: PTA Registry
Record Dates: First submitted 2016-02-18; First posted 2016-04-05 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Percutaneous Transluminal Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Percutaneous transluminal angioplasty (PTA) is a minimally invasive procedure for dilating blood vessels in the treatment of peripheral artery disease.

The aim of this registry is to collect prospectively and systematically clinical research data from patients undergoing PTA. This registry is an open-end observational study to assess the characteristics and outcomes in patients with undergoing PTA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PTA

Exclusion Criteria:

* < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PTA
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Patency rate | 6 months
Creatinine level | 2 Days after PTA

SECONDARY OUTCOMES:
Mortality | 30 days
Days of Hospitalization | 12 months
  Days of Hospitalization at 12 months
Ankle-Brachial Index | 6 months and 12 months
  Clinical Improvement measured by Ankle-Brachial Index
walking distance | 6 months and 12 months
  Clinical Improvement measured by walking distance
Restenosis rate | 12 months
  Percentage of patients with restenosis at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

REFERENCES:
- [Derived] Baasen S, Stern M, Wischmann P, Schremmer J, Sansone R, Spieker M, Wolff G, Bonner F, Quast C, Heiss C, Kelm M, Busch L. Endovascular Treatment of Flow-Limiting Iliofemoral Stenosis Improves Left Ventricular Diastolic Function in Patients With HFpEF by Reducing Aortic Pulsatile Load. Circ Heart Fail. 2024 Sep;17(9):e011258. doi: 10.1161/CIRCHEARTFAILURE.123.011258. Epub 2024 Sep 9. PMID 39247971
- [Derived] Busch L, Heinen Y, Stern M, Wolff G, Ozaslan G, Tzetou K, Sansone R, Heiss C, Kelm M. Angioplasty of Flow-Limiting Stenosis Reduces Aortic and Brachial Blood Pressure in Patients With Peripheral Artery Disease. J Am Heart Assoc. 2021 Jul 20;10(14):e019724. doi: 10.1161/JAHA.120.019724. Epub 2021 Jul 6. PMID 34227407